CLINICAL TRIAL: NCT06676176
Title: Psoriatic Arthritis Pathobiology and Its Relationship With Clinical Disease Activity
Acronym: PSABRE
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 010368 BHT
Record Dates: First submitted 2017-07-20; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: This study will be an observational study of a cohort of psoriatic arthritis patients who have failed to achieve sufficient response to standard non-biologic therapy. As they start their next treatment, this study aims to investigate the evolution of these patients in terms of the clinical, molecular and cellular profiles within the joint lining, peripheral blood and skin.

SUMMARY:
The study aims to examine the relationship between synovial histopathology and change in clinical disease activity over time in a population of patients with psoriatic arthritis who have failed to respond to first-line treatment. It is a prospective, open-labelled study

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 75 years of age inclusive;
2. Patients with Psoriatic Arthritis as defined by the CASPAR criteria;
3. Patients who have persistent active disease (defined as having 3 or more swollen and 3 or more tender joints) despite an adequate trial of 2 or more standard non-biologic disease-modifying drugs, administered either individually or in combination;
4. Subjects who are naïve to biologic therapy or who have experienced but failed one previous class of biologic agent;
5. The patient must be able to comply with the study visit schedule, treatment plans, lab tests and other study procedures;
6. The patient must be capable of giving informed consent.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding;
2. Men and women of childbearing potential who decline to employ adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) for the duration of the study;
3. As per care within a standard NHS setting, active infections of a serious nature such as HIV, HBV, pneumonia, or pyelonephritis are to be excluded. A history of previous serious infection is to be assessed individually for risk of re-activation, and a decision to treat (and with which agent) would be made according to the treating physician's discretion, as would normally occur within standard care. Less serious infections (such as upper respiratory tract infection [colds] or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator;
4. Active TB, or evidence of latent TB without adequate therapy for TB, initiated prior to first dose of biologic. Also excluded are patients with evidence of an old or latent TB infection without documented adequate therapy. Patients with previous or current close contact with an individual with active TB, or history of active TB, and patients who have completed treatment for active TB should have had a thorough evaluation for TB prior to study enrolment as recommended by a local infectious disease specialist or published local guidelines of TB control agencies;
5. History of septic arthritis within a native joint within the last 12 months;
6. Presence of a transplanted organ (with the exception of a corneal transplant occurring more than 3 months prior to screening);
7. Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated, with no evidence of recurrence);
8. History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly;
9. Known recent substance abuse (drug or alcohol);
10. History of or current primary inflammatory joint disease or primary rheumatological autoimmune disease other than PsA;
11. Poor tolerability of venepuncture required for blood sampling during the study period;
12. Patients unable to tolerate synovial biopsy or in whom this is contraindicated (e.g. on anti-coagulants may not be suitable). However, assessment of suitability for the biopsy procedure will be a local decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of PsA patients who have persistent disease activity despite an adequate trial of standard non-biologic disease-modifying therapy, and who may proceed to receive their first or second biologic drug as the next treatment strategy.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
DAS | 4 months
  The primary outcome measure is the Disease Activity Score (DAS), a composite score calculated using the Ritchie articular index (range 0-78), swollen joint count (range 0-44), patient--scored global health assessment on a visual analogue scale (range 0-100) and lab--measured erythrocyte sedimentation rate (ESR). This is used to assess the relationship between the level of interleukin(IL)-23 within the psoriatic arthritis synovium and clinical disease activity over time.

SECONDARY OUTCOMES:
Relationship between IL-23 levels within the PsA synovium/ skin and clinical disease activity | 4 months
Relationship between clinical disease activity and synovial, skin and/or blood levels of key immune signalling molecules involved in psoriatic disease | 4 months
  Such as but not limited to cluster of differentiation (CD)3, CD68, FVIII, TNFα, IL-1, IFN-γ, IL-6, IL-17A, IL-17R, IL-20, IL-22, IL-23/12p40, IL-23R, ICAM-1, VCAM-1, TGF-β, VEGF, PDGF, RANK-L, OPG, DKK-1, PNAd, CXCL13, CCL 21, MRP8 (S100A8), MRP14 (S100A9), Complement C3, TGFβ etc.
Relationship, if any, between clinical disease characteristics and genotype | 4 months
Relationship between activated inflammatory cells in psoriatic skin and those in the psoriatic synovium | 4 months
Relationship between clinical disease activity and synovitis, assessed using grey scale with power doppler US imaging | 4 months
Relationship between clinical enthesitis scores (eg. LEI) and US scores of enthesitis | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No